CLINICAL TRIAL: NCT06849986
Title: Tislelizumab Combined With Liposomal Doxorubicin and Ifosfamide as First-line Treatment for Patients With Specified Subtypes of Unresectable or Metastatic Soft Tissue Sarcoma: a Multi-center, Single-arm, Prospective Phase II Clinical Trial
Brief Title: IO Combined With AI as First-line Treatment for Patients With Soft Tissue Sarcoma(TAIS)
Acronym: TAIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2501312-5
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-03

CONDITIONS: Soft Tissue Sarcomas; Angiosarcoma; Fibrosarcoma; Leiomyosarcoma; Pleomorphic Liposarcoma; Malignant Peripheral Nerve Sheath Tumor (MPNST); Desmoplastic Small Round Cell Tumor
Keywords: soft tissue sarcoma; tislelizumab; doxorubicin; ifosfamide
MeSH Terms: conditions — Sarcoma; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Desmoplastic Small Round Cell Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- tislelizumab combined with AI (Experimental): Liposomal Doxorubicin (PLD) 30mg/m2 on day 1 Ifosfamide (IFO) 3 g/m2/day on days 1 to 3 Tislelizumab 200mg on day 1, administered by intravenous infusion, every 3 weeks
  Interventions: Drug: Tislelizumab+liposomal doxorubicin+ifosfamide

INTERVENTIONS:
Drug: Tislelizumab+liposomal doxorubicin+ifosfamide — Liposomal Doxorubicin (PLD) 30mg/m2 on day 1 Ifosfamide (IFO) 3 g/m2/day on days 1 to 3 Tislelizumab 200mg on day 1, administered by intravenous infusion, every 3 weeks

SUMMARY:
This study will enroll patients with specific subtypes of unresectable or metastatic soft tissue sarcoma, and will combine tislelizumab with the standard chemotherapy of liposomal doxorubicin and ifosfamide to initially explore the efficacy and safety.

DETAILED DESCRIPTION:
Soft tissue sarcoma is a type of malignant tumor originating from the mesenchymal tissue of soft tissues and visceral organs, and can occur in various parts of the human body. The incidence of soft tissue sarcoma accounts for about 1% of all adult malignant tumors and 15% of pediatric malignant tumors. Surgical resection is the cornerstone of soft tissue sarcoma treatment, but since soft tissue sarcomas often metastasize systemically, even early-stage cases can see lung metastasis. Except for solitary lung metastases, which still advocate surgical resection, the rest all require drug treatment, especially for the treatment of locally advanced or metastatic soft tissue sarcoma, systemic chemotherapy is the main means of clinical application.

Once soft tissue sarcoma metastasizes to a distant site, the prognosis is extremely poor, with a median survival time of less than 1 year. Clinical research results show that doxorubicin (ADM) is the basic and standard drug for the treatment of soft tissue sarcoma, and the combination of ADM and ifosfamide (IFO) (AI regimen) can increase the effective rate to 35%. The AI regimen is a commonly used first-line combination treatment for advanced soft tissue sarcoma.

Immune checkpoints have been approved by the FDA for the clinical treatment of various types of tumors. This study will enroll patients with specific subtypes of unresectable or metastatic soft tissue sarcoma, and will combine tislelizumab with the standard chemotherapy of liposomal doxorubicin and ifosfamide to initially explore the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years, regardless of gender;
* Patients with histopathologically confirmed undifferentiated sarcoma (except small round cell undifferentiated sarcoma), synovial sarcoma, angiosarcoma, fibrosarcoma, smooth muscle sarcoma, liposarcoma (except well differentiated liposarcoma), pleomorphic rhabdomyosarcoma, malignant peripheral nerve sheath meningiomas, desmoplastic small round cell tumor, not other specified (NOS), SMARCA4-deficient sarcoma, malignant phyllodes tumor of the breast, intimal sarcoma.
* Patients with locally advanced disease that is not amenable to surgery/radiation therapy or with recurrent/metastatic disease;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 to 1;
* Expected survival of more than 3 months;
* Within 7 days prior to screening (including day 7), laboratory test data requirements: neutrophil count ≥1.5×10⁹/L, platelet count ≥90×10⁹/L, hemoglobin ≥90g/L (no blood transfusion within 14 days), serum total bilirubin ≤1.5 times the upper limit of normal (ULN); ALT and AST ≤2.5× ULN (≤5× ULN for patients with liver metastases); serum creatinine ≤1.5× ULN or creatinine clearance rate ≥50ml/min;
* Presence of measurable lesions according to RECIST 1.1 criteria;
* The subject (or their legal representative/guardian) must sign an informed consent form, indicating that they understand the purpose of this study, are aware of the necessary procedures, and are willing to participate in this study.

Exclusion Criteria:

Any of the following conditions will result in exclusion from the study:

* Previous treatment for advanced soft tissue sarcoma, except for those who relapsed more than six months after adjuvant therapy with a cumulative dose of doxorubicin ≤300mg/m2;
* Received any experimental or anti - tumor drugs within 4 weeks prior to enrollment;
* Previously received any anti - PD - 1, anti - PD - L1, anti - PD - L2, anti - CD137, or anti - CTLA - 4 antibody treatment, or any other antibodies or drugs specifically targeting T - cell co - stimulation or checkpoint pathways;
* History of other tumors within the past five years, except for cured cervical cancer or skin basal cell carcinoma; for patients with post - radiation sarcoma, another primary tumor must have no recurrence or metastasis;
* Symptomatic brain or meningeal metastasis (unless the patient has been treated for more than 6 months, with negative imaging results within 4 weeks prior to enrollment, and stable tumor - related clinical symptoms at the time of enrollment);
* Clinically significant active bleeding;
* Pregnant or lactating women; women of childbearing potential who have not taken adequate contraceptive measures;
* Alcohol abuse or drug addiction;
* Patients with active autoimmune diseases or a history of such diseases that may recur (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.), or those at high risk (such as patients who have undergone organ transplantation and require immunosuppressive therapy). Autoimmune hypothyroidism requiring only hormone replacement therapy or skin diseases not requiring systemic treatment are excluded;
* Patients who need to receive systemic corticosteroids (equivalent to >10mg prednisone/day) within 14 days prior to enrollment or during the study, or those who require other immunosuppressive drug treatment. The use of topical or inhaled corticosteroids, or short - term (≤7 days) use of corticosteroids for prevention or treatment of non - autoimmune, non - frequent allergic diseases is excluded;
* Failure of important organs or other severe diseases, including interstitial pneumonia, clinically significant coronary artery disease, cardiovascular disease, or myocardial infarction, congestive heart failure, unstable angina, symptomatic pericardial effusion, or unstable arrhythmia within 6 months prior to enrollment;
* History of human immunodeficiency virus infection, or other acquired or congenital immune deficiency diseases, or history of organ transplantation or stem cell transplantation;
* Patients with active chronic hepatitis B or active hepatitis C. HBV carriers, those with stable hepatitis B after drug treatment (DNA titer ≤10^3 copies/ml), and those with cured hepatitis C (HCV RNA negative) are eligible for enrollment;
* Severe neurological or psychiatric history; severe infection; active disseminated intravascular coagulation, or other concomitant diseases that, in the opinion of the investigator, seriously endanger the safety of the patient or affect the patient's ability to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | Time from the date of recruiting to the first recorded complete remission (CR) or partial remission (PR), assessed up to 36 months.
  Defined as the percentage of participants in the analysis population who experienced a Complete Response or a Partial Response and was assessed using RECIST 1.1 based on investigator evaluation.

SECONDARY OUTCOMES:
PFS | From the date of recruiting to the date of first recorded progression or death from any cause, whichever comes first, assessed up to 36 months.
  Defined as the time from experiment drug administration to documented disease progression per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) or death due to any cause, whichever occurred first and was based on investigato evaluation.
OS | From recruiting to the time of death from any cause, assessed up to 36 months.
  Defined as the time from experiment drug administration to death due to any cause
Health Questionnaire Form | During the screening period, the second cycle and other even numbered cycles, each cycle is 21 days, assessed up to 36 months.
  Health Questionnaire Form

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Judson I, Verweij J, Gelderblom H, Hartmann JT, Schoffski P, Blay JY, Kerst JM, Sufliarsky J, Whelan J, Hohenberger P, Krarup-Hansen A, Alcindor T, Marreaud S, Litiere S, Hermans C, Fisher C, Hogendoorn PC, dei Tos AP, van der Graaf WT; European Organisation and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. Doxorubicin alone versus intensified doxorubicin plus ifosfamide for first-line treatment of advanced or metastatic soft-tissue sarcoma: a randomised controlled phase 3 trial. Lancet Oncol. 2014 Apr;15(4):415-23. doi: 10.1016/S1470-2045(14)70063-4. Epub 2014 Mar 5. PMID 24618336
- [Background] Shi Y, Su H, Song Y, Jiang W, Sun X, Qian W, Zhang W, Gao Y, Jin Z, Zhou J, Jin C, Zou L, Qiu L, Li W, Yang J, Hou M, Zeng S, Zhang Q, Hu J, Zhou H, Xiong Y, Liu P. Safety and activity of sintilimab in patients with relapsed or refractory classical Hodgkin lymphoma (ORIENT-1): a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2019 Jan;6(1):e12-e19. doi: 10.1016/S2352-3026(18)30192-3. PMID 30612710
- [Background] Tawbi HA, Burgess M, Bolejack V, Van Tine BA, Schuetze SM, Hu J, D'Angelo S, Attia S, Riedel RF, Priebat DA, Movva S, Davis LE, Okuno SH, Reed DR, Crowley J, Butterfield LH, Salazar R, Rodriguez-Canales J, Lazar AJ, Wistuba II, Baker LH, Maki RG, Reinke D, Patel S. Pembrolizumab in advanced soft-tissue sarcoma and bone sarcoma (SARC028): a multicentre, two-cohort, single-arm, open-label, phase 2 trial. Lancet Oncol. 2017 Nov;18(11):1493-1501. doi: 10.1016/S1470-2045(17)30624-1. Epub 2017 Oct 4. PMID 28988646